CLINICAL TRIAL: NCT06748170
Title: Al to Improve the Diagnosis of Rare Rheumatic Diseases
Acronym: AIDRARER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 24-221 ANZ
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Rheumatic Diseases
Keywords: Large language models; Diagnostic decision support; Clinical reasoning; rheumatology
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: The trial will be designed as a randomized, two-arm, single-blind parallel group study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Group will be given access to ChatGPT and standardized initial prompt
  Interventions: Other: ChatGPT
- Control group (No Intervention): Group will not be given access to any LLMs including ChatGPT but will be motivated to use other resources (such as online search enginges, Pubmed)

INTERVENTIONS:
Other: ChatGPT — OpenAI's ChatGPT language model with chat interface.
  Arms: Intervention group

SUMMARY:
This trial aims to assess the impact of providing medical students with access to ChatGPT, a state-of-the-art large language model, in comparison to conventional diagnostic decision support tools, on their diagnostic accuracy for rare rheumatic diseases.

DETAILED DESCRIPTION:
Advanced artificial intelligence (AI) technologies, particularly large language models such as OpenAI's ChatGPT, hold significant potential for enhancing medical decision-making. While ChatGPT was not specifically designed for medical applications, it has shown utility in various healthcare scenarios, including answering patient inquiries, drafting medical documentation, and aiding consultations. Despite these advancements, its role in supporting diagnostic reasoning-especially among less experienced medical students-and for complex rare diseases remains underexplored.

Diagnostic reasoning is a multifaceted process that combines pattern recognition, knowledge synthesis, and probabilistic thinking. Tools like ChatGPT could potentially alleviate cognitive burden, enhance diagnostic accuracy, and ultimately accelerate the diagnosis for rare diseases. However, ChatGPT is not tailored for diagnostic reasoning and lacks comprehensive validation in this domain. Additionally, it is susceptible to generating misinformation or plausible-sounding but inaccurate responses, which may hinder rather than support clinical decision-making. Therefore, understanding how medical students utilize such AI tools is essential before they are integrated into educational or clinical workflows. This study will also assess a standardized prompt to facilitate ChatGPT usage and will give students direct access to enable a realistic scenario.

This study will investigate the impact of ChatGPT on the diagnostic accuracy of medical students when tackling cases of rare rheumatic diseases. Participants will be randomized into two groups: one with access to ChatGPT and one using conventional diagnostic tools. Each participant will analyze diagnostic cases by providing up to 5 differential diagnoses and and rating the diagnostic confidence. Independent reviewers, blinded to group allocation, will evaluate the accuracy and quality of their responses. This study hence aims to provide insights into the potential benefits and limitations of integrating AI tools like ChatGPT.

ELIGIBILITY:
Inclusion Criteria:

* Medical students having started with clinical subjects (Internal medicine)

Exclusion Criteria:

* Not being a medical student

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of top diagnosis | during evaluation
  Participants in each group will make at least one disease suggestion (top diagnosis) and up to a total of a maximum of 5 suggestions. Percentage of exact matches of the top suggestion with the actual diagnosis will be analyzed

SECONDARY OUTCOMES:
Diagnostic accuracy of top 5 suggestions | during evaluation
  Participants in each group will make at least one disease suggestion (top diagnosis) and up to a total of a maximum of 5 suggestions. Percentage of exact matches with the actual diagnosis included in the top 5 suggestions will be analyzed
Diagnostic reasoning | during evaluation
  For each case, participants will receive 1 point for each plausible diagnosis and 2 points for a completely correct response. The total scores will be compared between the randomized groups.
Diagnostic confidence | during evaluation
  For each case participants will be asked for their diagnostic confidence (VAS 0-10). The mean score will be compared between groups.
Time spent for diagnosis | during evaluation
  We will compare how much time (in seconds) participants spend per case between the two study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Digital Medicine, University Hospital of Giessen and Marburg, Philipps University Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No